CLINICAL TRIAL: NCT06786455
Title: Pharmacokinetics, Pharmacodynamics, Safety, and Preliminary Efficacy of Subcutaneous Injection of SHR-1905 in Adolescent Asthmatic Subjects - an Open-label, Single-dose Phase II Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1905-204
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1905 Injection (Experimental)
  Interventions: Drug: SHR-1905 Injection

INTERVENTIONS:
Drug: SHR-1905 Injection — SHR-1905 Injection,medium dose, administered by subcutaneous injection;

SUMMARY:
Pharmacokinetics, pharmacodynamics, safety, and preliminary efficacy of subcutaneous injection of SHR-1905 in adolescent asthmatic subjects - an open-label, single-dose Phase II clinical study

ELIGIBILITY:
Inclusion Criteria:

1. The age of signing the informed consent must be ≥12 years old and <18 years old, both male and female.
2. Body weight ≥30 kg and BMI≥18 kg/m2.
3. The clinical diagnosis was asthma for at least 6 months.
4. Subjects receiving asthma maintenance therapy were required to maintain a stable dose for 4 weeks prior to baseline.
5. FEV1/ estimated value of pre-BD before bronchodilator in screening period must be ≥40%.
6. Screening period bronchial dilation test or bronchial excitation test positive.
7. Informed consent was signed before the trial.
8. Potentially fertile subjects voluntarily take appropriate contraceptive measures.

Exclusion Criteria:

1. Combined with clinically significant lung disease other than asthma
2. A combination of diseases other than asthma that may affect lung function
3. Combined with other pulmonary or systemic diseases associated with eosinophil elevation, or other diseases associated with eosinophil elevation that the investigators believe need to be excluded.
4. Bronchial thermoplasty or bronchial cryoablation were performed within 1 year prior to baseline.
5. Acute asthma attacks requiring systemic glucocorticoid use for ≥3 days occurred within 1 month prior to baseline.
6. Systemic glucocorticoids were used as maintenance therapy for the first 3 months of the baseline period.
7. Acute episodes of life-threatening asthma occurred within 5 years prior to baseline.
8. Allergen immunotherapy was administered 8 weeks prior to baseline.
9. Non-selective beta-blockers were used for the first 4 weeks of the baseline period.
10. Participated in clinical trials of any drug or medical device within 12 weeks prior to screening.
11. Severe trauma or major surgery in the 6 months prior to baseline.
12. History of malignant tumor.
13. Combined with serious other systemic diseases.
14. Combined with immunodeficiency disease.
15. A history of infection requiring treatment with systemic anti-infective drugs in the 4 weeks prior to baseline.
16. Parasitic infection was present in the 6 months prior to baseline.
17. Abnormal laboratory tests during screening or baseline. Screening or baseline ECG results were abnormal and clinically significant.
18. At the time of screening, smokers were still smoking or had quit for less than 6 months, or had a smoking history of ≥10 pack-years.
19. Alcohol consumption within 1 month prior to baseline.
20. History of drug abuse and drug use within 1 year before screening.
21. Those who had a history of blood donation within 4 weeks prior to baseline, or had significant blood loss, or had received a blood transfusion within 8 weeks.
22. People who received live (attenuated) vaccine or viral vector vaccine within 8 weeks prior to the baseline period or planned to receive it during the trial.
23. Researchers and relevant staff of research centres or others directly involved in programme implementation.
24. The investigator considers that there are any circumstances that may cause subjects to be unable to complete the study or present a significant risk to subjects or other factors that may reduce the likelihood of enrollment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
PK index: Serum SHR-1905 concentration。 | Day 253
PK index: Area under the plasma concentration versus time curve (AUC)。 | Day 253
PK index: Peak Plasma Concentration (Cmax）。 | Day 253
safety: Incidence and severity of any adverse events。 | Day 253

SECONDARY OUTCOMES:
PD index: Change of peripheral blood eosinophils absolute value (EOS) from baseline. | Day 253
Initial efficacy measures: Changes in forced expiratory volume in the first second (FEV1) from baseline. | Day 253
Initial efficacy measures: Changes in exhaled nitric oxide (FeNO) from baseline. | Day 253

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided